CLINICAL TRIAL: NCT04800250
Title: Mucogain Matrix Versus Connective Tissue Graft: "MUCOGREFFE Project"
Brief Title: Treatment of Multiple Gingival Recession Defects Using a New Xenogenic Collagen Membrane Compared to Connective Tissue Graft: a Randomized Controlled Split-mouth Clinical Study
Acronym: Mucogreffe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-PP-26
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Case-control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Mucogain matrix on right (Experimental): The patient will receive mucogain matrix on right side and connective tissue graft on left side.
  Interventions: Procedure: Treatment of gingival recessions
- B - Mucogain matrix on left (Experimental): The patient will receive mucogain matrix on left side and connective tissue graft on right side.
  Interventions: Procedure: Treatment of gingival recessions

INTERVENTIONS:
Procedure: Treatment of gingival recessions — Patients will have a surgery for their gingival recessions. They will be enrolled in the split mouth-study. They will have on one side mucogain matrix transplant, an on another side they will have the gold standard procedure

SUMMARY:
Limitation of donor site and significant postoperative morbidity are often described in connective tissue graft. We want to show if mucogain matrix used in tunnel technique to recover RTI Cairo recessions defects could be an alternative to connective tissue graft

ELIGIBILITY:
Inclusion criteria:

* Patient with 3 contiguous, symmetrical and bilateral RTI Cairo gingival recessions (Miller Class 1) (i.e. 6 recessions)
* Patient non-smoker
* Patient affiliated to social security
* Patient signed informed consent.

Exclusion criteria:

* Patient with or having presented an acute or chronic severe cardiovascular, kidney, liver, gastrointestinal, allergic, endocrine, neuropsychiatric pathology, developed cancer of the upper aero digestive tract treated with radiotherapy
* Patient with severe hemorrhinopathy
* Patient treated with oral retinoids, bisphosphonates, oral or anticonvulsants
* Patient who has taken steroidal or non-steroidal anti-inflammatory therapy, anti-cancer or immunosuppressive chemotherapy within the last 6 months.
* Patient with contraindication to necessary and pre-, per- or post-operative treatments
* Follow-up of the patient seemed difficult by the investigator
* Patient with insufficient oral hygiene incompatible with oral surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Mean root coverage obtained with both techniques | 6 months
  To compare the mean root coverage obtained with the Creos® Mucogain matrix and connective tissue graft in the treatment of Cairo RT1 class maxillary recessions (Miller Class 1).

SECONDARY OUTCOMES:
Postoperative pain with both techniques | 6 months
  To compare postoperative pain with both techniques
Postoperative complications with both techniques | 10 days
  To compare the occurrence of postoperative complications (haemorrhage, edema) within the first 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Provence-Alpes-Côte d'Azur Region, France

IPD SHARING:
Plan to Share IPD: No